CLINICAL TRIAL: NCT06811506
Title: Effect of Different Size of Patellar Resurfacing on Patellar Crepitus of the One-stage Bilateral Total Knee Arthroplasty: a Prospective Randomize Control Trial.
Brief Title: Effect of Different Size of Patellar Resurfacing on Patellar Crepitus of the One-stage Bilateral Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, piya pinsornsak, Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Patella crep TUH
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis (OA) of the Knee; OA Knee
Keywords: patella crepitation; crepitus; patella clunk
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Procedure: Anatomical size patella component
- Group 2 (Active Comparator)
  Interventions: Procedure: Reduced size patella component

INTERVENTIONS:
Procedure: Anatomical size patella component — After the patella was resurfaced, surgeon evaluated the symmetry through haptic feedback and assessed the thickness by measuring the distance from the anterior to posterior center of the patella. An inset, single pegged patella component was cemented after milling the patella. The patella was medialized as the patella bone would allow. Synovium laying on top of the femoral component with the knee in extension was routinely excised. Lateral facetectomy and restoration of native patella thickness were performed in all knees. In the control group, anatomically sized patella components were used.
  Arms: Group 1
Procedure: Reduced size patella component — The same procedure of patella resurfacing as control group was done, then 3 mm reduced size patella component was used in the intervention group.
  Arms: Group 2

SUMMARY:
The goal of this study is to compare the incidence of patella crepitation using different size of patella component in bilateral simultaneously total knee arthroplasty with patella resurfacing. The main question is does size of patella component effect the incidence of patella crepitus? In the control group, anatomically sized patella components were used, whereas the intervention group received 3 mm smaller, reduced-size patella components. Participants were scheduled for follow up examination 2 weeks, 6 weeks, 6 months and 1 year for incidence of the patella crepitation and other outcomes.

DETAILED DESCRIPTION:
For decades, total knee arthroplasty (TKA) has been the treatment of choice for knee osteoarthritis, with posterior-stabilized (PS) systems showing excellent long-term outcomes. However, patellar crepitus is more common with PS TKA systems because the cam and post mechanism can entrap fibrosynovial tissue within the intercondylar box, causing crepitus or clunking. Patellar crepitus (PC) was defined as an audible grinding noise or palpable vibrations in the knee during active and passive range of motion, detected by the examiner's hand on the patient's patella and sometimes can be audible.

This study was designed as a single-center, prospective randomized controlled trial comparing anatomical and reduced size of patella component in patients who underwent sequential bilateral TKA with patella resurfacing under single anesthesia. All participants were blinded to their intervention. A total of 94 knees from 47 patients were randomly assigned to undergo TKA with an anatomically sized patella component in one knee and reduced-size patella component in another knee or vice versa.

Crepitus, as a primary outcome, was assessed at 2, 6, 24 and 48 weeks follow-up using a validated and standardized approach. Crepitus was graded as: 0 (none), 1 (fine palpable), 2 (coarse palpable), and 3 (audible). Secondary outcomes included anterior knee pain (AKP), Feller's patella score (FPS), Kujala score, knee society score (KSS), range of motion (ROM), radiographic findings, and complications. AKP was measured using a 10-cm visual analog scale (VAS) in 1-cm increments. Knee ROM was measured with a goniometer. Radiographic parameters were measured at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80 years.
* American Society of Anesthesiologists (ASA) Classification 1 or 2.
* Diagnosed with primary knee osteoarthritis and requires bilateral total knee arthroplasty with patellar resurfacing.
* Participants can understand and consent to participate in the research project

Exclusion Criteria:

* Secondary knee osteoarthritis,
* Previous knee surgery or arthroscopic surgery
* Individuals who cannot undergo surgery due to underlying medical conditions.
* BMI > 40 kg/m2
* Infection around the knee

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patella crepitation | From postoperative follow-up 2 weeks to 1 year
  Crepitus was assessed at each follow-up using a validated and standardized approach of physical examination. The patient lay supine with relaxed muscles while the examiner passively flexed and extended the knee through a 30-90° range at least three times. Crepitus was graded as: 0 (none), 1 (fine palpable), 2 (coarse palpable), and 3 (audible).

SECONDARY OUTCOMES:
Range of motion | From enrollment (preoperative measurement) to the end of postoperative follow-up (1 year)
  Range of motion (flexion, extension) of the knee measure by long arm goniometer (record in degrees)
anterior knee pain | follow up 6 months and 12 months
  Define as pain originate from anterior aspect of the knee including patellofemoral joint especially when perform active range of motion of the knee. Measure in scale (0 means best, 10 means worst)
Feller's patella score | follow up 6 months and 12 months
  The questionnaire of Feller et al. [8] includes items on anterior knee pain, quadriceps strength, and ability to rise from a chair and climb stairs; these scores range from 3 to 30 points, with 30 points representing the best possible score.
Knee society score | follow up 6 months and 12 months
  1. "Knee Score" section (7 items) and a 2. "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Kujala score | follow up 6 months and 12 months
  13-item self-report questionnaire that assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. With 100 being the highest possible score. Lower scores reflect greater pain and disability.
Posterior tibial slope | preoperative and follow up 6 months
  The angle of the tibial plateau or tibial component from anterior to posterior relative to the longitudinal axis of the tibia. Measure in degrees on film true lateral knee flexion 30 degrees.
modified Patella tendon length | preoperative and follow up 6 months
  Measuring from the tibial tubercle's proximal point to the patella's distal articular facet. Measure in millimeters on film true lateral knee flexion 30 degrees.
modified Patella height | preoperative and follow up 6 months
  Measured from the distal to the proximal point of the same facet. Measure in millimeters on film true lateral knee flexion 30 degrees.
modified Insall salvati ratio | preoperative and follow up 6 months
  modified Insall-Salvati ratio = modified Patella tendon length / modified patella height
Posterior femoral offset | preoperative and follow up 6 months
  Defined as the maximum thickness of posterior condyle / femoral component projecting to the tangent of the posterior cortex of femoral shaft. Measure in millimeters on film true lateral knee flexion 30 degrees.
Patella tilt | preoperative and follow up 6 months
  The angle between the transverse axis of the patella and the anterior intercondylar line. Measure in degrees on film knee patella skyline.
Complication | up to 12 months
  Surgical site infection, deep infection or wound complication

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Nueng, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chumchuen S, Kanitnate S, Wattanasirisombat K, Tammachote N. Synovium removal from the articular side of the quadriceps tendon around the superior pole of patella reduces the crepitus after total knee arthroplasty. Int Orthop. 2022 Nov;46(11):2561-2567. doi: 10.1007/s00264-022-05539-2. Epub 2022 Aug 13. PMID 35962233
- [Background] Joseph L, Batailler C, Roger J, Swan J, Servien E, Lustig S. Patellar component size effects patellar tilt in total knee arthroplasty with patellar resurfacing. Knee Surg Sports Traumatol Arthrosc. 2021 Feb;29(2):553-562. doi: 10.1007/s00167-020-05984-9. Epub 2020 Apr 9. PMID 32274550
- [Background] Conrad DN, Dennis DA. Patellofemoral crepitus after total knee arthroplasty: etiology and preventive measures. Clin Orthop Surg. 2014 Mar;6(1):9-19. doi: 10.4055/cios.2014.6.1.9. Epub 2014 Feb 14. PMID 24605184
- [Background] Ogawa H, Matsumoto K, Akiyama H. Effect of Patellar Resurfacing on Patellofemoral Crepitus in Posterior-Stabilized Total Knee Arthroplasty. J Arthroplasty. 2016 Aug;31(8):1792-6. doi: 10.1016/j.arth.2016.01.023. Epub 2016 Jan 21. PMID 26948175
- [Background] Dennis DA, Kim RH, Johnson DR, Springer BD, Fehring TK, Sharma A. The John Insall Award: control-matched evaluation of painful patellar Crepitus after total knee arthroplasty. Clin Orthop Relat Res. 2011 Jan;469(1):10-7. doi: 10.1007/s11999-010-1485-3. PMID 20706813
- [Background] Thiengwittayaporn S, Sumranwanich N, Hongku N, Sansawat P. Onlay Patellar Resurfacing in a Posterior-Stabilized Total Knee Arthroplasty Increases Patellar Crepitus Complication: A Randomized, Controlled Trial. J Arthroplasty. 2021 Oct;36(10):3443-3450. doi: 10.1016/j.arth.2021.05.031. Epub 2021 May 27. PMID 34116913